CLINICAL TRIAL: NCT01562938
Title: A Phase 1, Randomized, Double-Blind, Placebo-controlled Study to Evaluate the Safety and Tolerability of MEDI-557, a Humanized Monoclonal Antibody With an Extended Half-life Against Respiratory Syncytial Virus (RSV), Administered to Healthy Adults
Brief Title: MEDI-557 Adult Dosing
Acronym: CD-1092
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: CD-ID-MEDI-557-1092
Record Dates: First submitted 2012-03-07; First posted 2012-03-26 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-10

CONDITIONS: Respiratory Syncytial Virus
Keywords: Respiratory Syncytial Virus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- MEDI-557 low-dose (Active Comparator)
  Interventions: Drug: MEDI-557
- MEDI-557 high-dose (Active Comparator)
  Interventions: Drug: MEDI-557

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: MEDI-557 — MEDI-557 low-dose
  Arms: MEDI-557 low-dose
Drug: MEDI-557 — MEDI-557 high-dose
  Arms: MEDI-557 high-dose

SUMMARY:
This is a Phase 1, double-blind, placebo controlled study enrolling 42 healthy adult subjects (18-45yrs) from 1 site. Subjects will be randomized in a 2:3:2 ratio to receive MEDI-557 or placebo. Subjects will receive 1 intravenous dose on Study Day 1. Subjects will be followed for safety from the time of Informed Consent through 360 days post dose.

DETAILED DESCRIPTION:
A Phase 1, randomized, double-blind, placebo-controlled study evaluating the safety and tolerability of MEDI-557 administered IV to healthy adult subjects (18-45yrs). A maximum of 42 subjects from 1 site will be enrolled in a 2:3:2 ratio (12 placebo, 18 MEDI-557 low-dose, 12 MEDI-557 high-dose) to allow for greater data collection in the low-dose group. Subjects are evaluated for safety from time of Informed Consent through Study Day 360 post dose.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* written informed consent obtained from subject prior to performing any protocol related procedures
* healthy by medical history and physical exam
* females of child-bearing potential must use 2 effective methods of birth control for 14 days prior to 1st dose and through 1 year after administration of study drug
* nonsterilized, sexually active males with female partner of child-bearing potential must use 2 effective methods of birth control from Day 1 through Day 361
* weight </= 110kg with a body mass index of <32kg/m2
* ability to complete a follow-up period of approximately 360 days

Exclusion Criteria:

* inability to complete a follow-up period of 360 days
* any condition in the opinion of investigator that would interfere with evaluation of IP or interpretation of subject safety or study results
* concurrent enrollment in another clinical study
* employees of the site or other individuals involved with the conduct of the study or immediate family members of such individuals
* receipt of immunoglobulin or blood products within 60 days prior to randomziation
* receipt of any investigational drug therapy within 6 months prior to IP dosing
* clinically abnormal ECG at screening
* blood donation in excess of 400mL, wihtin 6 months prior to randomization
* previous receipt fo biologics
* history of immunodeficiency
* history of allergic disease or reactions likely to be exacerbated by any component of the IP
* previous medical history or evidence of interurrent illness that may compromise the safety of the subject
* positive lab test for Hep A, B, C or HIV
* pregnancy or nursing mother
* history of alcohol or drug abuse within past 2 years
* positive urine Class A drug screen
* acute illness within 7 days prior to randomization
* fever >/= 99.5F witin 7 days prior to randomization
* any drug therapy within 7 days prior to randomization
* systolic BP >150mmHG and/or diastolic BP>90mmHg
* receipt of vaccine within 14 days prior to randomization
* abnormal study labs (hem/wbc/platelet/BUN - see protocol for specific information)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability | from time of informed consent through 360 days post dose (approximately 1 year total)
  The occurrence of AEs and SAEs
Safety and Tolerability | Pre-dose; every 30 minutes during infusion; up to 24 hours after end of infusion
  Vital sign measurements - blood pressure, heart rate, respiratory rate, temperature
Safety and Tolerability | from Day 1 (pre-dose) through 360 days post dose.
  Clinical lab measurements - chemistry, hematology; Urinalysis

SECONDARY OUTCOMES:
Pharmacokinetic Assessments - Serum | 1st dose through 360 days post dose
  Maximum serum concentration; Time to maximum serum concentration; Terminal phase elimination half-life; Area under the serum concentration-time curve from time zero to last measurable time point; Area under the serum concentration-time curve from time zero to infinity; Clearance; Volume of distribution
Occurrence of anti-MEDI-557 antibody - Serum and Nasal Wash | 1st dose through 360 days post dose
  MEDI-557 concentrations in serum and nasal wash through 360 days post dose
Pharmacokinetic Assessments - Nasal Wash | 1st dose through 360 days post dose
  Maximum nasal wash concentration; Time to maximum nasal wash concentration; Area under the nasal wash conentration-time curve from time zero to last measurable time point
anti-RSV antibody in Serum and Nasal Wash | 1st dose through 360 days post dose
  To evaluate anti-RSV antibodies (F-specific IgG and neutralizing) in serum and nasal wash.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Feldman, MD, Principal Investigator — Research Site; Hasan Jafri, Study Director — MedImmune LLC
Locations (1):
- Research Site, Miami, Florida, United States